CLINICAL TRIAL: NCT03687489
Title: Safety and Efficacy Study of Abdominal Aortic Aneurysm Stent Graft System for Infrarenal Abdominal Aortic Aneurysm: A Prospective, Multi-center, Objective Performance Criteria Clinical Trial
Brief Title: Safety and Efficacy Study of Abdominal Aortic Aneurysm Stent Graft System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lifetech Scientific (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTAAA-01
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm Stent Graft System
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Participants will be treated with Abdominal Aortic Aneurysm Stent Graft System
  Interventions: Device: Abdominal Aortic Aneurysm Stent Graft System

INTERVENTIONS:
Device: Abdominal Aortic Aneurysm Stent Graft System — Abdominal aortic bifurcation stent and iliac artery extension stent were preloaded into abdominal aortic bifurcation stent transporter and iliac artery extension stent transporter, respectively. In the operation, the abdominal aorta bifurcation stent and the iliac artery extension stent will be delivered to the corresponding lesion position of the abdominal iliac artery and release. The abdominal aortic bifurcation stent and the iliac artery extension stent will form a whole through docking and thereby reducing the risk of rupture of an infrarenal abdominal aortic aneurysm due to the shock of blood flow.

SUMMARY:
A prospective, multi-centre, objective performance criteria clinical trial to evaluate the safety and efficacy of Abdominal Aortic Aneurysm Stent Graft System manufactured by Lifetech Scientific (Shenzhen) Co., LTD. for the infrarenal abdominal aortic aneurysm.

DETAILED DESCRIPTION:
This clinical trial was conducted in a qualified clinical trial institution. Investigators will use Abdominal Aortic Aneurysm Stent Graft System manufactured by Lifetech Scientific (Shenzhen) Co., LTD. to treat patients with Infrarenal Abdominal Aortic Aneurysm. This is a Prospective, Multi-center, Objective Performance Criteria Clinical Trial. It is expected to submit to the ethics committee of the lead unit for review in March 2018, and complete the implantation of 156 patients in 22 centres nationwide within 12 months, and interim follow-up was conducted before discharge, 30 days after surgery, 6 months after surgery and 12 months after surgery, long-term follow-up will be performed at 24 months postoperatively, 36 months postoperatively, 48 months postoperatively and 60 months postoperatively.

This trial will evaluate whether the device reached the primary safety endpoint and primary efficacy endpoint through two primary endpoint indicators: the incidence of major adverse events (MAE) within 30 days and the success rate of abdominal aortic aneurysm treatment 12 months after surgery. This trail will evaluate whether the device reached the secondary safety endpoint and primary efficacy endpoint through several secondary endpoint indicators: Perioperative (intraoperative to postoperative 30 days) delivery related complications incidence rate (including the transabdominal surgery caused by intraoperative conveyors, the hemorrhage in the middle iliac artery, the hemorrhage in the femoral artery at the puncture site, the hematoma and the pseudoaneurysm), the incidence of acute lower limb ischemia before discharge and 30 days after surgery, all-cause mortality at 6 months, 12 months and 2-5 years after surgery, abdominal aortic aneurysm-related mortality at 6 months, 12 months and 2-5 years after surgery, the incidence of severe adverse events (SAE) at 6 months, 12 months and 2-5 years after surgery, the incidence of the device-related adverse events (AE) at 6 months, 12 months and 2-5 years after surgery, the incidence of type I or type III leakage at 6 months, 12 months after surgery, the incidence of displacement of Abdominal Aortic Aneurysm Stent at 6 months, 12 months after surgery and the incidence of conversion from abdominal aortic aneurysm treatment to open surgery or secondary surgery intervention at 6 months, 12 months and 2-5 years after surgery. According to the guidelines for clinical trials of aortic stent system, the sponsor will apply for CFDA listing registration after completing a 12-month primary endpoint assessment. According to the guidelines for clinical trials of aortic covered stent system, the sponsor will apply for CFDA listing registration after completing a 12-month primary endpoint assessment, and annually follow-up will be conducted until the fifth year for the long-term efficacy observation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged greater than 18 years old and less than 85 years old, regardless of gender.

  2. Patients who can understand the purpose of the trial, voluntarily participate in and sign the informed consent, and are willing to complete the follow-up according to the requirements of the protocol.

  3. Patients diagnosed with Infrarenal Abdominal Aortic Aneurysm and should meet at least one of the following conditions:
  1. The maximum diameter of abdominal aortic aneurysm ≥50mm in male patients, or the maximum diameter of abdominal aortic aneurysm ≥45mm in female patients.
  2. The maximum diameter of abdominal aortic aneurysm ≥40mm and the diameter increased by more than 5mm in the last 6 months (In this case, the diameter data of abdominal aortic aneurysm should be traceable within 6 months).
  3. The abdominal aortic aneurysm compresses vital organs and causes symptoms (such as abdominal pain, lower back pain, etc.) 4. The range of proximal aneurysm neck diameter of the abdominal aortic aneurysm is between 17mm to 32mm.

     5. The length of the proximal aneurysm neck of abdominal aortic aneurysm≥10mm, and the angle of the proximal aneurysm neck ≤75 °.

     6. The range of the diameter of the iliac artery anchoring area is between 8mm to 22mm.

     7.The length of the iliac artery anchoring area≥15mm.

     8. The patient has a suitable iliac and femoral artery approach.

     Exclusion Criteria:
* 1. Patients with severe stenosis, calcification, or mural thrombus in the anchoring area of the stent and easily lead to incomplete stent apposition.

  2. Patients with rupture of an abdominal aortic aneurysm or threatened rupture.

  3. Patients with abdominal aortic dissection.

  4. Patients with mycotic or infectious abdominal aortic aneurysms.

  5. Patients with a history of myocardial infarction or unstable angina pectoris for 6 months. Characteristics of unstable angina pectoris: angina symptoms gradually increased, new onset of rest or night angina pectoris or occurrence of angina prolonged.

  6. Patients with any transient ischemic attack (TIA) or ischemic stroke within 3 months.

  7. Patients with a history of allergy to contrast media, stents and conveyor materials (including nickel and titanium, polyester, PTFE, and nylon polymer materials).

  8. A patient with connective tissue diseases such as Marfan syndrome, Eaton syndrome, or Bessel's disease.

  9. Patients with liver dysfunction: Alanine transaminase (ALT) or Aspartate transaminase (AST) were five times higher than the normal upper limit；serum total bilirubin (STB) was two times higher than the normal upper limit.

  10. Patients with renal dysfunction: Serum creatinine (Cr) was two times higher than the normal upper limit.

  11. Life expectancy is less than one year.

  12. Patients with major organ failure or other serious diseases;

  13. Patients who were not suitable for endovascular treatment, judged by the investigator.

  14. Pregnant or lactating women or women who plan to get pregnant.

  15. The patients participated in other clinical trials and did not come out of the group or withdraw within the first 3 months of the screening period of this trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2020-11-30 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The success rate of abdominal aortic aneurysm treatment | 12 months after operation
  A successful abdominal aortic aneurysm treatment is a composite index and refers to the following criteria simultaneously:
  1. the immediate technical success (the immediate technical success refers to the delivery system is successfully delivered to a predetermined location, the abdominal aortic stent is successfully deployed, and the transporter can be safely withdrawn from the body).
  2. the increase of maximum diameter of abdominal aortic aneurysm at the 12th month after surgery ≤5mm, compared with that before surgery.
  3. The displacement of anterior abdominal aortic stent was no more than 10mm at the 12th month after the operation from the location before discharge.
  4. No type I or type III leakage requiring additional intervention occurred 12 months after surgery。 No abdominal aortic aneurysm rupture within 12 months after surgery.

SECONDARY OUTCOMES:
The incidence of Major Adverse Event (MAE) | 30 days after surgery
  Major Adverse Event (MAE) is defined as all-cause death, myocardial infarction, renal failure, respiratory failure, paraplegia, stroke, and intestinal ischemia.
Incidence of type I or III leakage | 6 months, 12 months after surgery
  Type I leakage is also known as peripheral leakage or graft related leakage, which refers to internal leakage resulting from the inability of stent-type blood vessels to adhere closely to an autologous blood vessel, and the blood flow continues to flow into the aneurysm cavity, including proximal type I and distal type I leakage. Type III leakage refers to leakage caused by the failure of stent-type vessels to bind themselves tightly or the rupture of artificial vessels, and the blood flow continues to flow into the aneurysm cavity.
The incidence of abdominal aortic stent displacement | 6 months, 12 months after surgery
  The displacement refers to the position of abdominal aorta stents of postoperative follow-up are displaced more than 10 mm from the before discharge position.
Operation efficacy - incidence of conversion from abdominal aortic aneurysm treatment to open surgery or secondary surgery | 6 months, 12 months and 2-5 years after surgery.
  The incidence of conversion from abdominal aortic aneurysm treatment to open surgery or secondary surgery intervention.
The incidence rate of perioperative delivery related complications | intraoperative and postoperative 30 days.
  Perioperative period refers to intraoperative time to 30 days postoperative. Delivery related complications incidence including he transabdominal surgery caused by intraoperative conveyors, the hemorrhage in the middle iliac artery, the hemorrhage in the femoral artery at the puncture site, the hematoma and the pseudoaneurysm.
The incidence of Acute lower limb ischemia. | Before discharge and 30 days after surgery
  The incidence of acute lower limb ischemia.
All-cause mortality | 6 months, 12 months and 2-5 years after surgery
  All-cause mortality evaluates at 6 months, 12 months and 2-5 years after surgery
Disease related mortality | 6 months, 12 months and 2-5 years after surgery
  Abdominal aortic aneurysm-related mortality evaluates at 6 months, 12 months and 2-5 years after surgery.
Severe adverse events (SAE) | 6 months, 12 months and 2-5 years after surgery
  The incidence of severe adverse events (SAE). According to the ISO 14155 SAE refers to
  1. led to death,
  2. led to serious deterioration in the health of the subject, that either resulted in
     1. a life-threatening illness or injury, or
     2. a permanent impairment of a body structure or a body function, or
     3. in-patient or prolonged hospitalization, or
     4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function,
  3. led to foetal distress, foetal death or a congenital abnormality or birth defect
Device-related adverse effects (AE) | 6 months, 12 months and 2-5 years after surgery
  The incidence of the device-related adverse effects (AE), according to the ISO14155, adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Professor, Principal Investigator — Chinese PLA General Hospita
Locations (22):
- China (22):
  - Chinese PLA General Hospita, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The Frist Hospital of Lanzhou University, Lanzhou, Gansu
  - Liuzhou General Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Second Hospital of Heibei Medical University, Shijiazhuang, Hebei
  - Renming Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shanghai Ninth People's Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Xijing Hospital, The Fourth Military Medical University, Xi’an, Shanxi
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Tianjing Medical University General Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Frist Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Yan'an Hospital of Kunming City, Kunming, Yunnan
  - The Frist Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang